CLINICAL TRIAL: NCT01894399
Title: Phase I Study to Assess the Safety, Tolerability, Pharmacokinetic Characteristics of HM61713 Tablet in Healthy Korean, Japanese and Caucasian
Brief Title: Study to Evaluate a Pharmacokinetic of HM61713 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMSI-102
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
Keywords: HM61713; pharmacokinetics; Phase I; healthy; olmutinib
MeSH Terms: interventions — olmutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental): 100 mg HM61713 single dose in Korean
  Interventions: Drug: HM61713
- Cohort 2 (Experimental): 200 mg HM61713 single dose in Korean
  Interventions: Drug: HM61713
- Cohort 3 (Experimental): 300 mg HM61713 single dose in Korean
  Interventions: Drug: HM61713
- Cohort 4 (Experimental): 200 mg HM61713 single dose in Japanese
  Interventions: Drug: HM61713
- Cohort 5 (Experimental): 300 mg HM61713 single dose in Japanese
  Interventions: Drug: HM61713
- Cohort 6 (Experimental): 200 mg HM61713 single dose in Caucasian
  Interventions: Drug: HM61713
- Cohort 7 (Experimental): 300 mg HM61713 single dose in Caucasian
  Interventions: Drug: HM61713

INTERVENTIONS:
Drug: HM61713 — Cohort 1 : 100mg single dose in Korean Cohort 2 : 200mg single dose in Korean Cohort 3 : 300mg single dose in Korean Cohort 4 : 200mg single dose in Japanese Cohort 5 : 300mg single dose in Japanese Cohort 6 : 200mg single dose in Caucasian Cohort 7 : 300mg single dose in Caucasian
  Other Names: Olmutinib

SUMMARY:
Study Design

* Open, escalating single-dose design.
* 7 ascending dose cohorts
* In each cohorts, subjects will receive a single dose of HM61713.
* Main objective of this study is to evaluate the pharmacokinetics of HM61713 tablet.

DETAILED DESCRIPTION:
Primary objectives

• To assess the PK characteristics of HM61713 and metabolites in healthy male volunteers

Secondary objectives

* To assess the safety and tolerability of HM61713 tablet in healthy male subjects.
* To assess the food effect on PK characteristics of HM61713 tablet in healthy male subjects.
* To assess the ethnic differences of PK characteristics of HM61713 (Korean, Japanese, Caucasian)
* To investigate genotype of drug metabolism.transport that affect PK characteristics of HM61713
* To investigate the change of endogenous metabolic markers after administration of HM61713

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 20 and 45
* Informed of the investigational nature of this study and voluntarily agree to participate in this study
* BMI of >18.5kg/m2 and <28kg/m2 subject

Exclusion Criteria:

* Use of any prescription medication within 2 weeks prior to Day 1
* Use of any medication within 1 weeks prior to Day 1
* Has a severe medical history of hypersensitivity to drug
* Participation in another clinical study within 8 weeks days prior to start of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of HM61713 and metabolites | 0-48 hrs
Area under the plasma concentration time curve from zero to infinity (AUC) of HM61713 and metabolites | 0-48 hrs
Tmax of HM61713 and metabolites | 0-48 hrs
Terminal half life (t1/2) of HM61713 and metabolites | 0-48 hrs
The apparent plasma clearance (CL/F) of HM61713 and metabolites | 0-48 hrs
Mean residence time (MRT) of HM61713 and metabolites | 0-48 hrs

SECONDARY OUTCOMES:
Safety data, including physical examinations, laboratory evaluation, ECGs, ICGs, vital signs, and adverse events. | 7 days after the investigational drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Research Site, Seoul, South Korea